CLINICAL TRIAL: NCT01662271
Title: Course of Obesity and Extreme Obesity in Adolescents, in the Context of Different Treatment Options - a Longitudinal Prospective Observation Study
Brief Title: Course of Obesity and Extreme Obesity in Adolescents
Acronym: YES
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Martin Wabitsch (Other)
Collaborators: University of Witten/Herdecke (Other); Charite University, Berlin, Germany (Other); University of Leipzig (Other); Universität Duisburg-Essen (Other); Helmholtz Zentrum München (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. Martin Wabitsch, Division Chief Pediatric Endocrinology and Diabetology, University of Ulm
Organization: University of Ulm (Other)
Other Study IDs: U1111-1131-4384e; DRKS00004172 (Registry Identifier: Deutsches Register Klinischer Studien); 01GI1120A (Other Grant/Funding Number: Bundesministerium für Bildung und Forschung)
Record Dates: First submitted 2012-07-20; First posted 2012-08-10 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Obesity; Extreme Obesity
Keywords: obesity; adiposity; psychosocial; healthcare; co-morbidities; youth with extreme obesity; weight loss
MeSH Terms: conditions — Obesity; Obesity, Morbid; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of fasting plasma, serum, DNA, and urine will be retained.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- adolescents with extreme obesity: BMI ≥35kg/m2
- adolescents with obesity: BMI 30-34.9kg/m2

SUMMARY:
The rate of adolescent extreme obesity is rapidly rising, and impacting quality of life, psychosocial situation, and health of the affected youth. However, as few of these adolescents seek medical care, little is known about the longitudinal course of adolescent extreme obesity.

In this study, the investigators aim to provide structured care for adolescents with obesity and extreme obesity over a prolonged period of time, and to gain information on the course of obesity and the success of different treatment options. The study is a subproject of the "Medical and psychosocial implications of adolescent extreme obesity - acceptance and effects of structured care", short: "Youth with Extreme obesity Study (YES)", which aims at improving the medical care and social support structures for youth with obesity and extreme obesity in Germany. Obese youth and young adults (BMI ≥ 30kg/m2) between the ages of 14 and 24.9 years (initially up to 21 years) are eligible to participate. Participants will have a physical check-up every 12 months (initially every 6 months), complete questionnaires on their health, socioeconomic status and wellbeing, and are offered blood test and diagnostic procedures to assess comorbidities. Participants are offered support and guidance for social and vocational integration. The study will evaluate and inform treatment and support options for adolescents with extreme obesity.

DETAILED DESCRIPTION:
Little is known about the longitudinal course of adolescent extreme obesity. In this multicenter study, the investigators aim to enroll adolescents with extreme obesity (BMI ≥ 35kg/m2) in a 9 year longitudinal, prospective observation that will reveal information on the course of obesity and the success of different treatment options. Adolescents with more moderate degrees of obesity (BMI 30-34,9kg/m2) will serve as a control group. The project builds on the Consortium "Medical and psychosocial implications of adolescent extreme obesity - acceptance and effects of structured care", short: "Youth with extreme obesity Study (YES)", which comprises the recruitment and characterization of obese youth from different healthcare- and non healthcare settings, a randomized controlled trial to investigate a novel intervention targeted at improving quality of life and social functioning of extremely obese adolescents, a structured prospective evaluation of adolescent bariatric surgery, and economic assessments of the financial burden of extreme adolescent obesity on the healthcare system.

Based on the current state of knowledge, the investigators have formulated the following a priori hypotheses in regards to the longitudinal observation study:

1. Youth with extreme obesity (BMI ≥ 35kg/m2) achieve lower adherence with the structured care program compared to adolescents with more moderate degrees of obesity (BMI 30-34,9kg/m2).
2. Youth with extreme obesity (BMI ≥ 35kg/m2) are less likely to achieve and sustain weight loss over a prolonged period of time, compared to adolescents with more moderate degrees of obesity (BMI 30-34,9kg/m2).
3. Youth with extreme obesity (BMI ≥ 35kg/m2) are harder to integrate in the job market compared to youth with more moderate degrees of obesity (BMI 30-34,9kg/m2).
4. Youth with extreme obesity (BMI ≥ 35kg/m2) have higher incidence and severity of co-morbidities compared to youth with more moderate degrees of obesity (BMI 30-34,9kg/m2).

The investigators aim to recruit a total of 600 adolescents age 14 to 24.9 years (initial age up to 21 years; changed in an amendment in February 2013) with extreme obesity (BMI ≥ 35 kg/m2) and 600 adolescents with obesity (BMI 30-34.9 kg/m2) over a 24 months period. The five participating university centers are distributed across 4 geographic regions in the North (Berlin), in the West (Essen/Datteln), in the East (Leipzig) and in the South (Ulm) of Germany, and will therefore render data that are representative of Germany as a whole. Adolescent will be examined annually (initially examinations were biannually, this was changed in an amendment in December 2014), and testing will include an array of standardized questionnaires and validated instruments to assess health, psycho-social situation, psychiatric co-morbidities and health related quality of life, as well as a physical examination, laboratory tests, and screenings for orthopedic co-morbidities and sleep apnea. Participants are offered support and guidance in regards to social and vocational integration with the aim of improving self esteem and social functioning. Data will be entered in an extended version of the "German National Register for Longitudinal Research on Childhood Obesity". We will perform sub-analyses based on the treatment options these youths have followed The project will reveal the acceptance and outcomes of a structured healthcare program for adolescents with extreme obesity and provide unique information on the medical and psychosocial development of adolescents with extreme obesity in Germany.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30kg/m2
* sufficient German language skills

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects will be recruited from the general population through different healthcare- and non healthcare settings to ascertain the inclusion of treatment-seeking and non treatment-seeking individuals. Healthcare settings include university based obesity clinics, physician offices and health insurance agencies. Non-healthcare settings include schools, job centers, and employment agencies.
Sampling Method: Non-Probability Sample
Enrollment: 429 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2023-07 (Actual); Study Completion 2023-07 (Actual)

PRIMARY OUTCOMES:
adherence with structured care | 12 months after subject inclusion
  The percentage of subjects that comply with the structured follow up program will be calculated once a year.

SECONDARY OUTCOMES:
percentage of subjects that can be integrated into the job-market or into an apprenticeship training position | every 12 months for 9 years
  The percentage of subjects who can be integrated into the job-market or into an apprenticeship training position will be determined via standardized questionnaire (modified after KIGGS and TeenLABS).
percentage of subjects that undergo the recommended diagnostic procedures | every 12 months for 9 years
  Medically appropriate diagnostic procedures will be recommended to the patients, and the percentage of subjects that undergo the recommended diagnostic procedures will be documented.
changes in somatic co-morbidities | every 12 months for 9 years
  Incidences and changes of somatic co-morbidities will be assessed via standardized physical examination, laboratory and apparative tests, and standardized patient questionnaires (modified after KIGGS and TeenLABS).
changes in psychiatric co-morbidities | every 12 months for 9 years
  Incidences and changes of psychiatric co-morbidities will be assessed via validated patient questionnaires once a year.
compliance with treatment of somatic co-morbidities | every 12 months for 9 years
  Appropriate treatment of the diagnosed somatic co-morbidities will be offered to all subjects. The percentage of subjects who comply with such therapy will be assessed via standardized questionnaire (modified after KIGGS and TeenLABS).
compliance with treatment of psychiatric co-morbidities | every 12 months for 9 years
  Appropriate treatment of the diagnosed psychiatric co-morbidities will be offered to all subjects. The percentage of subjects who comply with such therapy will be assessed via standardized questionnaire (modified after KIGGS and TeenLABS).
changes in health related quality of life | every 12 months for 9 years
  Assessed via validated questionnaires (EQ5D, DISABKIDS).
changes in socio-economic status | every 12 months for 9 years
  Assessed via standardized questionnaires (modified after KIGGS and TeenLABS).
incidence of extreme obesity | every 12 months for 9 years
  The incidence of extreme obesity (BMI ≥35kg/m2) will be determined in the group of adolescents with moderate obesity (BMI 30-34.9kg/m2).
changes in BMI-SDS | every 12 months for 9 years
  Height and weight will be measured with standardized instruments and BMI-SDS will be calculated.
predictors of the above outcomes | every 12 months for 9 years
  Psycho-social, psychiatric, and medical variables will be assessed via standardized physical examination, laboratory and apparative tests, standardized patient questionnaires (modified after KIGGS and TeenLABS), and validated psychiatric instruments once a year, and correlation with the outcome variable will be assessed via multiple regression analyses.
adherence with structured care | every 12 months from 2-9 years post enrollment
  The percentage of subjects that comply with the structured follow up program will be calculated once a year.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wabitsch, Prof. Dr. med., Study Chair — University of Ulm; Susanna Wiegand, Dr. med., Principal Investigator — Charite University, Berlin, Germany; Thomas Reinehr, Prof. Dr. med., Principal Investigator — University of Witten/Herdecke; Johannes Hebebrand, Prof. Dr. med., Principal Investigator — Universität Duisburg-Essen; Wieland Kiess, Prof. Dr. med., Principal Investigator — University of Leipzig; Reinhard Holl, Prof. Dr. med., Principal Investigator — University of Ulm
Locations (5):
- Germany (5):
  - Ambulatory Obesity Program, Charité University, Berlin, Berlin
  - Vestische Kinderklinik, University of Witten/Herdecke, Datteln
  - University Duisburg-Essen, Essen
  - University Hospital Leipzig, Leipzig
  - Dept for Pediatrics and Adolescent Medicine, University of Ulm: Interdisciplinary obesity clinic, Ulm

REFERENCES:
- [Derived] Wabitsch M, Moss A, Reinehr T, Wiegand S, Kiess W, Scherag A, Holl R, Holle R, Hebebrand J. Medical and psychosocial implications of adolescent extreme obesity - acceptance and effects of structured care, short: Youth with Extreme Obesity Study (YES). BMC Public Health. 2013 Aug 29;13:789. doi: 10.1186/1471-2458-13-789. PMID 23987123
- See also: study homepage — http://www.adipositasforschung-ulm.de/index.php?id=69